CLINICAL TRIAL: NCT01063387
Title: Molecular Markers in Lymph Node Metastasis of Cervical Cancer and Prophylactic Irradiation of the Para-Aortic Lymph Nodes and Supraclavicular Lymph Nodes in Locally Advanced Uterine Cervical Cancer
Brief Title: Prophylactic Irradiation of the Para-Aortic Lymph Nodes and Supraclavicular Lymph Nodes in Locally Advanced Uterine Cervical Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Ding Ma, Cancer Biology Research Center of Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GM2010-022
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2010-02-05 (Estimated); Status verified 2010-02

CONDITIONS: Cervical Cancer
Keywords: cervical cancer,semaphorin 4C (Sema4C),; Prophylactic Irradiation
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sema4c positive +Common iliac lymph nodes control (No Intervention): Sema4c Positive & "Radical hysterectomy +Pelvic Radiotherapy "
- Sema4c positive +Common iliac lymph nodes Experimental (Active Comparator): Sema4c Positive & "Radical hysterectomy+ EFI(whole pelvis + para-aortic lymph node irradiation) "
  Interventions: Radiation: Prophylactic Irradiation of the Para-Aortic Lymph Nodes and supraclavicular lymph nodes in Locally Advanced Uterine Cervical Cancer
- Sema4c Positive + PAN positive control arm (No Intervention): Sema4c Positive & " Radical hysterectomy+ EFI(whole pelvis + para-aortic lymph node irradiation) "
- Sema4c positive+ PAN positive Experimental (Experimental): Sema4c Positive & Radical hysterectomy+ EFI(whole pelvis + para-aortic lymph node irradiation+ supraclavicular lymph nodes irradiation) '
  Interventions: Radiation: Prophylactic Irradiation of the Para-Aortic Lymph Nodes and supraclavicular lymph nodes in Locally Advanced Uterine Cervical Cancer

INTERVENTIONS:
Radiation: Prophylactic Irradiation of the Para-Aortic Lymph Nodes and supraclavicular lymph nodes in Locally Advanced Uterine Cervical Cancer — Sema4c positive+ Para-aortic lymph node metastasis Experimental : Radiation: Extended-field Irradiation (EFI) Prophylactic irradiation of supraclavicular lymph node
  Arms: Sema4c positive+ PAN positive Experimental
Radiation: Prophylactic Irradiation of the Para-Aortic Lymph Nodes and supraclavicular lymph nodes in Locally Advanced Uterine Cervical Cancer — Sema4c positive +Common iliac lymph nodes metastasis Experimental :Radical hysterectomy+ EFI(whole pelvis + para-aortic lymph node irradiation)
  Arms: Sema4c positive +Common iliac lymph nodes Experimental

SUMMARY:
This study is an open-label, randomized study, which is designed to investigate the efficacy of Extended-field irradiation (EFI) on reducing recurrences at the para-aortic lymph node (PAN) and supraclavicular lymph nodes, and also on improving disease-free survival of locally advanced uterine cervical cancer. This study includes a translational research component in that all the primary tumors and lymph node are stained with Sema4c, before randomization. According to the investigators study result, patients with more pelvic lymph node metastasis are more likely to develop distant metastasis including the recurrences at PAN and supraclavicular lymph node. Primary cervical cancer tissues and lymph nodes are examined for expression of Sema4c just after registration, and before the patients are randomized to each arm (pelvis only vs. EFI). The investigators expect a higher benefit of EFI in patients with Sema4c-positive lymph node.

ELIGIBILITY:
Inclusion Criteria:

* Patients (who have been adequately clinically staged) with primary, untreated, histologically confirmed invasive squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the uterine cervix, FIGO stage IB1 with pelvic lymph node metastasis, IB2, IIA(≥4cm in tumor size, or pelvic LN metastasis), IIB, IIIA, IIIB? with only unilateral pelvic wall extension
* Patients with negative, para-aortic lymphadenopathy determined by pelvic MRI and/or PET/CT scan.
* Patients with adequate bone marrow function: ANC greater than or equal to 1,500/ul, platelets greater than or equal to 100,000/ul at the beginning.
* Patients with adequate renal function: creatinine equal to or less than 2.0 mg/dL.
* Patients who have signed an approved informed consent and authorization
* Patients with ECOG Performance Status of 0, 1, 2 and Karnofsky Performance Scale of 100, 90, 80, 70, 60, 50
* Age: 18≤age≤80

Exclusion Criteria:

* Stage IIIb with bilateral pelvic wall extension and stage IVB lesions are not eligible.
* Patients with histology other than squamous, adeno, adenosquamous cell carcinoma
* Patients who have received prior radiotherapy of pelvis or total hysterectomy Patients who have diagnosis of other malignant tumors other than non-malignant melanoma skin cancer or stage I. II papillary, follicular thyroid cancer.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2010-01; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of the Extended-Field Irradiation on the recurrence rate in para-aortic lymph nodes, supraclavicular lymph nodes and the disease-free survival rate of the patients with locally advanced uterine cervical cancer | 5 years

SECONDARY OUTCOMES:
To evaluate overall survival, toxicities and quality of life (QOL) of the patients treated by EFI compared to the control group of patients | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ma Ding, M.D., Study Director — Tongji Hospital of HUST
Locations (1):
- Tongji Hospital of HUST, Wuhan, Hubei, China